CLINICAL TRIAL: NCT04908228
Title: Fixed-duration Therapy With Ibrutinib and Obinutuzumab (GA-101) in Treatment-naïve Patients With CLL
Acronym: FIGHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paolo Ghia (Other)
Responsible Party: Sponsor-Investigator, Paolo Ghia, Prof, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-CLL-008
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibrutinib + obinutuzumab (Experimental): Ibrutinib 420 mg QD for 24 months (Cycles 1-24) Obinutuzumab starting from Cycle 13 Day 1 (100 mg Cycle 13 Day 1, 900 mg Cycle 13 Day 2, 1000 mg Cycle 13 Days 8 and 15, 1000 mg Cycles 14-18 Day 1).
  Interventions: Drug: Ibrutinib and obinutuzumab

INTERVENTIONS:
Drug: Ibrutinib and obinutuzumab — Patients will receive fixed-duration treatment with ibrutinib and obinutuzumab.
  Other Names: Imbruvica and Gazyvaro

SUMMARY:
This is a phase 2 multicenter national interventional pharmacological study aimed at determining the efficacy of a fixed duration treatment with ibrutinib and obinutuzumab in terms of uMRD in the BM at the end of treatment (+30 Days follow-up).

Treatment with ibrutinib and obinutuzumab will be administered according to the following schedule:

Ibrutinib 420 mg QD for 24 months (Cycles 1-24) Obinutuzumab starting from Cycle 13 Day 1 (100 mg Cycle 13 Day 1, 900 mg Cycle 13 Day 2, 1000 mg Cycle 13 Days 8 and 15, 1000 mg Cycles 14-18 Day 1).

At the end of Cycle 24 all responding patients will discontinue ibrutinib and proceed with follow-up. If disease relapse occurs at any time after discontinuing treatment, ibrutinib therapy will be reintroduced at the standard dose of 420 mg QD and response to treatment monitored over time. Patients with stable (SD) or progressive disease (PD) at the end of Cycle 24, will continue ibrutinib as long as the treating physician deems they are benefiting from treatment and will be followed up in the study for survival and response to subsequent therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that meets iwCLL diagnostic criteria
3. Previously untreated active disease requiring treatment per iwCLL criteria
4. ECOG PS 0 or 1
5. Measurable lymph node disease (>1.5 cm longest diameter) by CT scan
6. Adequate hematologic function defined as:

   1. Absolute neutrophil count (ANC) >750 cells/μL (750 cells/mm3 or 0.75 x 109/L)
   2. Platelet count >30,000/μL (30,000 cells/mm3 or 30 x 109/L)
   3. Hemoglobin >8.0 g/dL
7. Adequate hepatic and renal function defined as:

   1. Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤3.0 x upper limit of normal (ULN)
   2. Estimated Creatinine Clearance (CrCl) ≥30 mL/min (Cockcroft- Gault)
   3. Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
8. Prothrombin time (PT)/International normal ratio (INR) <1.5 x ULN and PTT (activated partial thromboplastin time [aPTT]) <1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder).

Exclusion Criteria:

Any prior therapy (including but not limited to chemotherapy, targeted therapy, immunomodulating therapy, radiotherapy, and/or monoclonal antibody) used for treatment of CLL or SLL.

2. Patients carrying del(17p) and/or TP53 mutation as assessed by central laboratory.

3. History of other malignancies, except:

1. Malignancy treated with curative intent and with no known active disease present for ≥3 before the first dose of study drug and felt to be at low risk for recurrence by the treating physician
2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
3. Adequately treated carcinoma in situ without evidence of disease. 4. Known or suspected history of Richter's transformation. 5. Known hypersensitivity to one or more study drugs. 6. Known bleeding disorders (eg, von Willebrand's disease or hemophilia). 7. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.

   8. Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrolment. Those who are PCR positive will be excluded. 9. Unable to swallow capsules/tablets or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.

   10. Concomitant use of warfarin or other vitamin K antagonists. 11. Major surgery within 4 weeks of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
BM MRD <10-4 at 30 days follow-up | 24 months
  To evaluate the rate of bone marrow minimal residual disease <10-4 at +30 Days follow-up after ibrutinib and obinutuzumab

SECONDARY OUTCOMES:
Overall response rate at 30 days follow-up | 24 months
  To evaluate response to treatment after ibrutinib and obinutuzumab

CONTACTS AND LOCATIONS:
Locations (1):
- Strategic Research Program on CLL, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No